CLINICAL TRIAL: NCT03317756
Title: CONfident Treatment Decisions in Living With Rheumatoid Arthritis
Acronym: CONTROL-RA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Pfizer Independent Grants for Learning and Change (Unknown)
Responsible Party: Principal Investigator, Maria Danila, MD, MSc, MSPH, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: X151222003
Record Dates: First submitted 2017-09-12; First posted 2017-10-23 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Masking Description: intervention and control arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Variation 1 (Experimental): Patient Educational Intervention: Patient will receive intervention videos and will be required to complete the baseline and follow-up surveys.
  Interventions: Other: Patient Educational Intervention
- Patient Variation 2 (Experimental): Patient Control: Patients will receive an attention control and will be required to complete the baseline and follow-up surveys.
  Interventions: Other: Patient Control

INTERVENTIONS:
Other: Patient Educational Intervention — Patients will view 5-6 videos that will help them with pre-identified patient barriers to achieving RA low disease activity
  Arms: Patient Variation 1
Other: Patient Control — Patients will receive an attention control
  Arms: Patient Variation 2

SUMMARY:
Pilot test the novel educational patient-directed intervention to demonstrate the feasibility of the novel educational approaches developed in improving patient's willingness to achieve remission or low disease activity in RA.

DETAILED DESCRIPTION:
Pilot test the novel educational patient-directed intervention to demonstrate the feasibility of the novel educational approaches developed in improving patient's willingness to achieve remission or low disease activity in RA. Upon agreement to participate, the patient participants will provide information on their treating physician. This information will be used to invite physicians to complete the physician-educational intervention and offered CME credits for completing the activity.

The investigators will recruit participants from a patient registry (1:1 intervention: control) that meet the eligibility criteria. The recruited patients will complete the educational intervention (if randomized to the intervention arm) and the study outcomes will be collected immediately after the intervention and also after the patients most proximate rheumatologist visit (up to 6-months later).

ELIGIBILITY:
Inclusion Criteria:

* Have a patient-reported diagnosis of RA
* Most recent RAPID3 > 12 collected in the last 6 months
* Have not changed RA medication in the last 6 months
* Taking medications that are commonly used in RA (e.g. methotrexate, sulfasalazine, hydroxychloroquine (plaquenil), leflunomide (arava), etanercept (enbrel), adalimumab (Humira), tofacitinib (xeljanz), actemra (tocilizumab), sarilumab (Kevzara) , infliximab (remicade), golimumab (Simponi), rituximab (rituxan), abatacept (Orencia), and certolizumab (Cimzia))

Exclusion Criteria:

* Does not meet inclusion criteria
* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Patient willingness to adopt T2T and the attainment of the T2T goals. | Follow-up Survey #1 (after completion of the intervention)
  Name of Scale: Choice predisposition scale The scale measures the willingness to change medication. The scale is a 11-point likert type scale that is scored from not willing at all (minimum) to extremely willing (maximum) with an unsure option (neutral).
  Higher scores (closer to the maximum) indicate a willingness to change medication and desire to further improve their RA disease activity.

OTHER OUTCOMES:
Acceptability of the educational interventions | Follow up Survey #1 (after completion of intervention)
  We will ask participants to rate the educational content.

CONTACTS AND LOCATIONS:
Overall Officials: Maria I Danila, MD MSc MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
No individual data. Aggregate results will be reported.